CLINICAL TRIAL: NCT04602026
Title: Re-Defining Frailty and Improving Outcomes Through Prehabilitation (RIOT Trial)
Brief Title: The RIOT Trial: Re-Defining Frailty and Improving Outcomes With Prehabilitation for Pancreatic, Liver, or Gastric Cancer
Acronym: RIOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Mark Rubinstein, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OSU-20057; NCI-2020-04925 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Adult Liver Carcinoma; Gastric Carcinoma; Malignant Solid Neoplasm; Pancreatic Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular; Stomach Neoplasms; Pancreatic Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (physical therapy consultation, exercise intervention) (Experimental): Patients undergo a physical therapy consultation and complete home exercises 3 days per week.
  Interventions: Behavioral: Exercise Intervention; Procedure: Physical Therapy; Other: Questionnaire Administration
- Arm II (best practice) (Active Comparator): Patients receive standard of care.
  Interventions: Other: Best Practice; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive standard of care
  Other Names: standard of care; standard therapy
  Arms: Arm II (best practice)
Behavioral: Exercise Intervention — Complete home exercise intervention
  Arms: Arm I (physical therapy consultation, exercise intervention)
Procedure: Physical Therapy — Undergo physical therapy
  Other Names: Physiatric Procedure; Physical Medicine Procedure; Physical Therapeutics; Physical Therapy Procedure; Physiotherapy; Physiotherapy Procedure; PT
  Arms: Arm I (physical therapy consultation, exercise intervention)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies how well a prehabilitation program works to improve patient outcomes after surgery compared to the normal standard of care prehabilitation in frail patients undergoing surgery for pancreatic, liver, or gastric cancer. Frailty is defined as the pathophysiology of aging or through the accumulation of physiologic and functional deficits. Prehabilitation programs seek to optimize the medical and physical state of patients prior to undergoing surgery with the goal of improving outcomes following surgery. Despite evidence for its importance in health outcomes for frail patients, prehabilitation programs have not been well studied in cancer surgery populations. This trial may provide researchers with more information on how to improve patient outcomes after cancer surgery through the use of prehabilitation programs.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To develop a novel, multi-dimensional index of physiologic reserve and resilience specific to surgical cancer patients.

II. To implement and assess a novel comprehensive multidimensional prehabilitation program on frail cancer surgery patients.

OUTLINE: All patients enrolled (both frail and non-frail) will be randomized (1:1) at the time of enrollment to receive pre-operative exercise or non-preoperative exercises. Randomization will be stratified by frailty status.

ARM I: Enrolled patients undergo a physical therapy consultation and complete home exercises 3 days per week, in addition to standard guidelines.

ARM II: Enrolled patients follow standard guidelines.

All patients are followed up at 2 weeks after surgery and then every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for any abdominal (e.g., pancreatic, liver or gastric) cancer surgery or established in the GI surgical oncology clinics or
* Scheduled for neoadjuvant therapy prior with the plan to be scheduled for surgery

Exclusion Criteria:

* Non-English speaking
* Prisoners
* Persons unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2024-12-09 (Actual)

PRIMARY OUTCOMES:
Frailty assessment | Baseline
  A rapid assessment for frailty using the widely used 5-item fatigue, resistance, ambulation, illness, & loss of weight (FRAIL) questionnaire will be performed. Patients are identified as frail by scoring 2 or more points on the FRAIL questionnaire. The frailty assessment will be aimed at identifying factors related to the 6 characteristics of frailty: physical performance, gait speed, mobility, nutritional status, mental health and cognition.
Morbidity | Baseline
  Will be assessed using standardized case report forms.
Complication burden | Baseline
  Will be calculated using the Comprehensive Complication Index (CCI). This method is more powerful than standard binary measures of morbidity (presence/absence of individual events) as it presents a quantitative score based on an aggregate weighted total ranging from 0 (no complications) to 100 (death).
Health-related quality of life (composite measure) | Baseline, 2 weeks, 3, 6, 12 months
  Will be recorded by administration of the Patient Reported Outcomes Measurement Information System (PROMIS) health-related quality of life questionnaire. PROMIS is a validated set of patient-centered measures that evaluates and monitors life domains (physical, mental, social health) and provide standardized patient reported outcome resources for use in clinical research and practice.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Rubinstein, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamad A, Zhang H, Zhang Y, Shen C, Fa P, Huang H, Ejaz A, Tsung A. Understanding the mechanism behind preoperative exercise therapy in patients with gastrointestinal cancers: a prospective randomized clinical trial. BMC Sports Sci Med Rehabil. 2025 Mar 14;17(1):50. doi: 10.1186/s13102-025-01094-6. PMID 40087747
- See also: The Jamesline — http://cancer.osu.edu

DOCUMENTS (1):
  • Informed Consent Form (2023-05-30): https://cdn.clinicaltrials.gov/large-docs/26/NCT04602026/ICF_000.pdf